CLINICAL TRIAL: NCT06744140
Title: Role of MRI Breast in Detection of Ductal Carcinoma in Situ
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHS/Batch-Spring23/018
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Carcinoma in Situ
MeSH Terms: conditions — Carcinoma in Situ | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging (MRI) — To Evaluate the breast Magnetic Resonance Imaging (MRI) in detecting Ductal Carcinoma In Situ (DCIS) lesions among high-risk breast cancer patients while keeping the histopathology as a GOLD standard

SUMMARY:
"This study investigates the role of Magnetic Resonance Imaging (MRI) in detecting Ductal Carcinoma in situ (DCIS) in high-risk breast cancer patients.

DETAILED DESCRIPTION:
Improved detection rates of DCIS in high-risk patients. Enhanced diagnostic accuracy, reducing false positives and negatives. Ductal Carcinoma in situ (DCIS) is a non-invasive breast cancer where abnormal cells are confined to the milk ducts.

The Breast Imaging Reporting and Data System (BI-RADS) is a standardized scoring system used to classify breast imaging findings. Scores range from 0 (incomplete) to 6 (known biopsy-proven malignancy)."

ELIGIBILITY:
Inclusion Criteria:

* High-risk breast cancer patients with a family history of breast cancer or genetic predispositions (e.g., BRCA mutations).
* Patients aged 30-65 years.
* Patients willing to undergo breast MRI screening for DCIS detection.

Exclusion Criteria:

* Patients with contraindications to MRI imaging (e.g., pacemakers, claustrophobia).
* Patients with a history of prior breast surgery or interventions that may interfere with imaging interpretation.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To Evaluate the breast Magnetic Resonance Imaging (MRI) in detecting Ductal Carcinoma In Situ (DCIS) lesions among high-risk breast cancer patients while keeping the histopathology as a GOLD standard
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-03-21 (Estimated)

PRIMARY OUTCOMES:
sensitivity & specificity | 12 Months
  sensitivity & specificity of MRI in detecting DCIS
BIRADS scores | 12 Months
  BIRADS scores will be used to evaluate the diagnostic accuracy of MRI in detecting DCIS

CONTACTS AND LOCATIONS:
Locations (1):
- INMOL hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No